CLINICAL TRIAL: NCT01129193
Title: Phase I Study of AR-42 in Relapsed Myeloma, Chronic Lymphocytic Leukemia, and Lymphoma
Brief Title: AR-42 in Treating Patients With Advanced or Relapsed Multiple Myeloma, Chronic Lymphocytic Leukemia, or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amir Mortazavi (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Arno Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Amir Mortazavi, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-09102; NCI-2010-01082 (Registry Identifier: Clinical Trials Reporting Program (CTRP)); P30CA016058 (NIH)
Record Dates: First submitted 2010-05-17; First posted 2010-05-24 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Prolymphocytic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Multiple Myeloma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Testicular Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Leukemia, Prolymphocytic; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Hematologic Malignancies) (Experimental): Patients will receive orally administered AR-42 three times per week (Mon, Wed, and Fri preferred) in cycles of 28 days (3 weeks of 3-times-per-week dosing followed by a 7-day off-treatment period).
  Interventions: Other: Pharmacodynamic Studies; Other: Fatigue Inventory; Other: Pharmacogenomic studies; Drug: AR-42
- Arm II (Solid Tumors) (Experimental): Patients will receive orally administered AR-42 three times per week (Mon, Wed, and Fri preferred) in cycles of 28 days (3 weeks of 3-times-per-week dosing followed by a 7-day off-treatment period).
  Interventions: Drug: AR-42

INTERVENTIONS:
Other: Pharmacodynamic Studies — Assess at baseline (pre-dose day 1 of cycle 1), approximately 24 hours after the first dose, pre-dose days 2 and 3, and pre-dose day 19 for histone acetylation of tumor cells (CLL patients) or mononuclear cells (PBMCs for lymphoma, myeloma, and solid tumor patients).
  Cytokine studies will be collected pre-dose on days 1, 2, 8, 15, 19 of cycle 1, day 1 of cycle 2, and pre-dose days 1, 8, 15 of cycle 3.
  Other Names: correlative studies
  Arms: Arm I (Hematologic Malignancies)
Other: Fatigue Inventory — Brief Fatigue Inventory should take each patient approximately 5 minutes to fill out this survey per instance on day 1 of every cycle.
  Other Names: quality-of-life assessmentBrief
  Arms: Arm I (Hematologic Malignancies)
Other: Pharmacogenomic studies — Baseline germ line DNA from buccal swabs will be collected for analysis of drug (AR-42) metabolism SNPs and other biologic SNPs that might predict immune or disease response to therapy. Pharmacogenetic status of key metabolizing enzymes (eg, CYP3A5, UGT1A8) and transporter proteins (SLCO1B1, ABCG2) will also be considered for their role in drug clearance in individual patients.
  Arms: Arm I (Hematologic Malignancies)
Drug: AR-42 — Administered orally three times per week (Mon, Wed, and Fri preferred) in cycles of 28 days (3 weeks of 3-times-per-week dosing followed by a 7-day off-treatment period).

SUMMARY:
RATIONALE: AR-42 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of AR-42 in treating patients with advanced or relapsed multiple myeloma, chronic lymphocytic leukemia, or lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the safety by estimating the maximum tolerated dose (MTD) and describe the dose limiting toxicity (DLT) of AR-42 administered orally three times weekly (Mon, Wed, and Fri preferred) each week for 3 weeks during each 28-day period to adults with advanced or recurrent chronic lymphocytic leukemia (CLL), lymphoma, or multiple myeloma (MM).

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetics of AR-42 in this patient population. II. To analyze patient samples for descriptive information regarding AR-42 pharmacodynamic changes in this patient population.

III. To obtain pilot data regarding efficacy at the MTD as measured by partial and complete responses in each disease subgroup during protocol expansion in stage III.

OUTLINE:

Patients receive oral AR-42 three times weekly on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 30 days.

ELIGIBILITY:
Inclusion Hematologic Malignances Arm

* Patients must have CLL, prolymphocytic leukemia, or lymphoma (Hodgkins or Non-Hodgkins) as defined by 2008 WHO criteria or multiple myeloma as defined by IMWG criteria
* Patients must have received at least one prior antineoplastic therapy, must have progressed after at least 1 prior therapy, and for whom no standard therapy is available or whom decline such options; prior autologous and/or allogeneic transplant is permitted
* Prior biologic therapy or prior radiation is permitted; however, at least 28 days must have elapsed since the completion of prior therapy and patients must have recovered from all therapy-associated toxicities to no greater than grade 1 at the time of registration
* Patients with symptomatic disease may receive palliative corticosteroids up to 1 week before initiating therapy
* Patients must be off any prior chemotherapy for at least 28 days or 3 half lives, whichever is longer, and all therapy-related toxicity must have resolved to grade 1 or less
* ANC >= 1000/uL
* Total bilirubin < 1.5 mg/dL
* Serum creatinine =< 1.5x institutional upper limit of normal or estimated creatinine clearance >= 50 ml/min by MDRD (original or abbreviated), or measured creatinine clearance >= 50 mL/min
* ECOG/WHO performance score of 0-1
* Patients must be able to swallow capsules
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial
* Women with potential for child bearing must have a negative pregnancy test at screening; both men and women are required to use appropriate contraception during study
* Platelet count >= 50,000/uL
* AST and ALT =< 5x the institutional upper limit of normal Inclusion Solid Tumors Arm
* Histologically or cytologically confirmed advanced or recurrent solid tumor malignancy.
* Chemotherapy: up to three prior cytotoxic chemotherapy treatments.
* Radiation Therapy: prior radiation therapy allowed.
* Surgery: Prior curative and palliative intent surgery is allowed.
* Age ≥ 18 years
* ECOG performance status 0-1
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below:
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin < 1.5 mg/dL
* AST(SGOT)/ALT(SGPT) ≤ 2.5 x institutional upper limit of normal (ULN); ≤ 5 x ULN in presence of liver metastasis
* Creatinine ≤ 1.5 x ULN OR Creatinine clearance ≥ 50 mL/min by MDRD (original or abbreviated), or measured creatinine clearance ≥ 50 ml/min
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial
* Women with potential for child bearing must have a negative pregnancy test at screening; both men and women are required to use appropriate contraception during study

Exclusion Hematologic Malignances Arm

* Pregnant women are excluded from this study
* Patients with malabsorption or any other condition that in the opinion of the principal investigator could cause difficulty in absorption of drug
* Breastfeeding should be discontinued if the mother is treated with AR-42
* Patients with malignant cells in the cerebrospinal fluid or parenchyma within the preceding 3 months or patients with primary CNS lymphoma are not eligible
* Patients with uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP) are not eligible
* Patients receiving concurrent corticosteroids less than 1 week prior to protocol therapy other than for physiologic maintenance treatment or control of AIHA or ITP
* Concurrent use of complementary or alternative medicines that in the opinion of the principal investigator would confound the interpretation of toxicities and/or antitumor activity of the study drug
* Patients with a "currently active" second malignancy that, in the opinion of the principal investigator, will interfere with patient participation, increase patient risk, shorten survival to < 1 year, or confound data interpretation
* Patients with a mean QTcB > 450 msec in males and > 470 msec in females
* Patients who are receiving concurrent antineoplastic therapy
* Any other medical condition, including mental illness or substance abuse, deemed by the principal investigator to likely interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results
* Patients with significant cardiovascular disease, including a myocardial infarction or unstable angina within 6 months or unstable cardiac arrhythmias are not eligible for the study
* Known HIV infection

Exclusion Solid Tumors Arm

* Pregnant women are excluded from this study
* Patients with malabsorption or any other condition that in the opinion of the principal investigator could cause difficulty in absorption of drug
* Patients with malignant cells in the cerebrospinal fluid or parenchyma within the preceding 3 months or patients with primary CNS lymphoma are not eligible
* Patients with uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP) are not eligible
* Patients receiving concurrent corticosteroids less than 1 week prior to protocol therapy other than for physiologic maintenance treatment or control of AIHA or ITP
* Concurrent use of complementary or alternative medicines that in the opinion of the principal investigator would confound the interpretation of toxicities and/or antitumor activity of the study drug
* Concurrent use of complementary or alternative medicines that in the opinion of the principal investigator would confound the interpretation of toxicities and/or antitumor activity of the study drug
* Patients with a "currently active" second malignancy that, in the opinion of the principal investigator, will interfere with patient participation, increase patient risk, shorten survival to < 1 year, or confound data interpretation.
* Patients with a mean QTcB > 450 msec in males and > 470 msec in females
* Patients who are receiving concurrent antineoplastic therapy.
* Any other medical condition, including mental illness or substance abuse, deemed by the principal investigator to likely interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* Patients with significant cardiovascular disease, including a myocardial infarction or unstable angina within 6 months or unstable cardiac arrhythmias are not eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-05-04 (Actual); Primary Completion 2017-01-07 (Actual); Study Completion 2017-01-07 (Actual)

PRIMARY OUTCOMES:
Adverse events described using the NCI CTCAE criteria | Up to 3 years

SECONDARY OUTCOMES:
Clinical benefit | Up to 3 years
Duration of response | Up to 3 years
Time to progression | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Amir Mortazavi, MD, Principal Investigator — The Ohio State University James Cancer Hospital
Locations (1):
- The Ohio State University James Cancer Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Collier KA, Valencia H, Newton H, Hade EM, Sborov DW, Cavaliere R, Poi M, Phelps MA, Liva SG, Coss CC, Wang J, Khountham S, Monk P, Shapiro CL, Piekarz R, Hofmeister CC, Welling DB, Mortazavi A. A phase 1 trial of the histone deacetylase inhibitor AR-42 in patients with neurofibromatosis type 2-associated tumors and advanced solid malignancies. Cancer Chemother Pharmacol. 2021 May;87(5):599-611. doi: 10.1007/s00280-020-04229-3. Epub 2021 Jan 25. PMID 33492438
- [Derived] Sborov DW, Canella A, Hade EM, Mo X, Khountham S, Wang J, Ni W, Poi M, Coss C, Liu Z, Phelps MA, Mortazavi A, Andritsos L, Baiocchi RA, Christian BA, Benson DM, Flynn J, Porcu P, Byrd JC, Pichiorri F, Hofmeister CC. A phase 1 trial of the HDAC inhibitor AR-42 in patients with multiple myeloma and T- and B-cell lymphomas. Leuk Lymphoma. 2017 Oct;58(10):2310-2318. doi: 10.1080/10428194.2017.1298751. Epub 2017 Mar 7. PMID 28270022
- [Derived] Cheng H, Xie Z, Jones WP, Wei XT, Liu Z, Wang D, Kulp SK, Wang J, Coss CC, Chen CS, Marcucci G, Garzon R, Covey JM, Phelps MA, Chan KK. Preclinical Pharmacokinetics Study of R- and S-Enantiomers of the Histone Deacetylase Inhibitor, AR-42 (NSC 731438), in Rodents. AAPS J. 2016 May;18(3):737-45. doi: 10.1208/s12248-016-9876-3. Epub 2016 Mar 4. PMID 26943915
- See also: The Jamesline — http://cancer.osu.edu